CLINICAL TRIAL: NCT06610240
Title: Perioperative Treatment Patterns and Clinical Outcomes in Early-Stage Non-Small Cell Lung Cancer: a Real-World Observational Study
Brief Title: Perioperative Treatment Outcomes of Early NSCLC
Acronym: Peri-R
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Hua Zhong, professor, Shanghai Chest Hospital
Other Study IDs: IS24118
Record Dates: First submitted 2024-09-11; First posted 2024-09-24 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: NSCLC
Keywords: NSCLC；; perioperative treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational study evaluating the clinical characteristics, treatment patterns, and clinical outcomes of perioperative NSCLC patients receiving different treatment strategies. According to the inclusion and exclusion criteria, perioperative NSCLC patients admitted to the study center from January 1, 2020, to one year after the study initiation will be retrospectively screened and collected.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III NSCLC patients confirmed by histological or cytological examination based on the 8th edition of the AJCC staging system.
* Patients who have undergone radical lung cancer surgery.
* Patients who have received neoadjuvant treatment before radical lung cancer surgery, including chemotherapy, targeted therapy, or immunotherapy both alone or combined.

Exclusion Criteria:

* Patients with other previous malignancies, except those who achieved complete remission at least two years before radical lung cancer surgery and did not require additional treatment.
* Patients with incomplete key baseline and treatment information，including clinical stage, pathological type, neoadjuvant treatment, pathological response, imaging response after neoadjuvant.
* Patients included in anti-tumor drug intervention or unblinded clinical trials, in which the treatment being administered is unknown.
* Prior surgery, radiotherapy or systemic therapy for NSCLC, including radiofrequency ablation, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: stage I-III NSCLC under different perioperative treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
event-free survival | From date of diagnosis until the date of first documented progression, recurrence or date of death from any cause, whichever came first, assessed up to 36 months
  the time from randomization to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause;
overall survival | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 60 months
  from diagnosis to death

SECONDARY OUTCOMES:
R0 resection rate | usually 1 week after surgery
  margin negative resection
major pathological response | usually 1 week after surgery
  viable tumor cell less than 10%
p-CR | usually 1 week after surgery
  no viable tumor cells was observed

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Dr., MD, Study Chair — Shanghai Chest Hospital
Locations (1):
- Zhong Hua, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
we need to further analyze the data